CLINICAL TRIAL: NCT01551706
Title: A Randomized, Double-blind, Placebo-controlled, Pilot Study to Evaluate the Effect of ENI Patented Whole Grape Extract on Antioxidant Status
Brief Title: Pilot Study to Evaluate the Effect of ENI Patented Whole Grape Extract on Antioxidant Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ethical Naturals, Inc. (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11OAHE
Record Dates: First submitted 2012-02-21; First posted 2012-03-13 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: High Oxidation Stress; Oxidized LDL Level
Keywords: Total antioxidant capacity; SOD; 8-OHdG; 8-isoprostane; oxLDL
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENI Patented Whole Grape Extract (Active Comparator): ENI Patented Whole Grape Extract (350 mg) per day
  Interventions: Dietary Supplement: ENI Patented Whole Grape Extract
- Exicipient pill (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ENI Patented Whole Grape Extract — ENI Patented Whole Grape Extract
  Other Names: Whole Grape Extract
  Arms: ENI Patented Whole Grape Extract
Other: Placebo — Placebo
  Other Names: Other ingredients pill
  Arms: Exicipient pill

SUMMARY:
This is a Randomized, Double-blind, Placebo-controlled, Pilot Study to Evaluate the Effect of ENI Patented Whole Grape Extract on Antioxidant Status.

DETAILED DESCRIPTION:
This study will investigate the effect of ENI Patented Whole Grape Extract versus placebo on antioxidant status. The primary objective is to determine antioxidant status by measuring total antioxidant capacity and superoxide dismutase (SOD) in blood and 8-OHdG and 8-isoprostane in first morning void urine samples prior to and after six weeks of supplementation with ENI Patented Whole Grape Extract.

Secondary objectives will include the assessment of oxidized LDL (oxLDL) and safety evaluations:

1. oxLDL
2. Safety laboratory tests: CBC, electrolytes, glucose, creatinine, eGFR, AST, ALT, GGT,bilirubin
3. Vital signs: heart rate and blood pressure
4. Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 - 65 years of age
2. If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

   OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Double-barrier method (condoms with spermicide or diaphragm with spermicide)
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Intrauterine devices
   * Vasectomy of partner (shown successful as per appropriate follow-up)
   * Abstinence
3. One or more of the following conditions:

   * Pre-hypertension defined as diastolic blood pressure of 80-89 mmHg and systolic blood pressure of 139 or lower at screening
   * BMI from 25.0 to 34.9 kg/m2
   * Pre-diabetes defined as a fasting plasma glucose from 5.2 to 6.9 mmol/L
4. Subjects who are smokers agree to report smoking habits at each visit and do not plan on changing their smoking habits during the study.
5. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Subject has any clinically significant medical conditions including cardiovascular disease,hypertension (systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90mmHg), diabetes, liver or kidney disease
3. Use of medication for the treatment of hypertension
4. Use of medication for vasodilation, including nitric oxide releasing patches
5. Use of medication for erectile dysfunction
6. Use of medication (prescribed or over the counter) for weight loss
7. Use of statins, fibrates, niacin, or any other medication for the treatment of hypercholesterolemia
8. Use of anticoagulants
9. Use of illicit drugs or history of drug or alcohol abuse with the past 5 years (currently having more than 2 standard alcoholic drinks per day)
10. Use of natural health products (NHPs)/dietary supplements that are known to have significant antioxidant activity within 2 weeks prior to baseline and during the course of the study including but not limited to vitamins A, C, and E, selenium and zinc.
11. Participation in a clinical research trial within 30 days prior to baseline
12. Clinically significant abnormal laboratory results at screening including

    * AST, ALT and/or bilirubin > 2 x the ULN
    * Serum creatinine >1.5 x the ULN or eGFR < 60
    * hemoglobin < 140 g/L for males and < 123 g/L for females
13. Allergy or sensitivity to test product ingredients
14. Individuals who are cognitively impaired and/or who are unable to give informed consent
15. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline on oxidation stress biomarkers including total antioxidant capacity, superoxide dismutase (SOD), 8-OHdG and 8-isoprostane | 6 weeks
  This study will investigate the effect of ENI Patented Whole Grape Extract versus placebo on antioxidant status. The primary objective is to determine antioxidant status by measuring total antioxidant capacity and superoxide dismutase (SOD) in blood and 8-OHdG and 8-isoprostane in first morning void urine samples prior to and after six weeks of supplementation with ENI Patented Whole Grape Extract.

SECONDARY OUTCOMES:
Change from baseline in oxidized LDL (oxLDL). | 6 weeks
  Secondary objectives will include the assessment of oxidized LDL (oxLDL)
Change from baseline in safety lab test biomarkers including CBC, electrolytes, glucose, creatinine, eGFR, AST, ALT, GGT, and bilirubin | 6 weeks
  This study will include the safety evaluations and measure if there are any abnormal levels of CBC, electrolytes, glucose, creatinine, eGFR, AST, ALT, GGT,and bilirubin.
Change from baseline in vital signs: heart rate and blood pressure | 6 weeks
  This study will include measurement on change from baseline in vital signs: heart rate and blood pressure
Number of participants with adverse events | 6 weeks
  This study will also assess number of participants with adverse events during the entire intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada